CLINICAL TRIAL: NCT02098707
Title: Effects of a Multidisciplinary Intensive Rehabilitation Treatment (MIRT) on Balance in Patients With Parkinson's Disease Evaluated With a Stabilometric Platform
Brief Title: Effects of a Rehabilitation Treatment on Balance in PD Evaluated With a Stabilometric Platform
Acronym: SPPD002
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Other Study IDs: SP PD 002; SPPD002 (Other: Ospedale generale di Zona "Moriggia-Pelascini")
Record Dates: First submitted 2014-03-21; First posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Parkinson Disease
Keywords: Stabilometric Platform; Rehabilitation; Balance Disorders; Falls
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 30 Parkinson disease patients: 30 patients (12 M, 18 F, mean age 66,8 ± 8,7) diagnosed with PD in stage 3 of Hoen&Yahr (mean Unified Parkinson Disease Rating Scale [UPDRS] III 18.8±10.5) will undergo a balance training using a stabilometric platform.
  Interventions: Other: Stabilometric Platform

INTERVENTIONS:
Other: Stabilometric Platform — Stabilometric platform is a device used for assessment and training of balance basing on ground reaction force evaluation in static conditions.

SUMMARY:
Pharmacotherapy with dopaminergic medications and deep brain stimulation cannot provide significant improvements in postural instability in Parkinson's disease, whereas previous reports of physical interventions have suggested promising results. The investigators want to study the effects of the multidisciplinary intensive rehabilitation treatment (MIRT) on balance disorders in Parkinson Disease (PD).

DETAILED DESCRIPTION:
Pharmacotherapy with dopaminergic medications and deep brain stimulation cannot provide significant improvements in postural instability in Parkinson's disease, whereas previous reports of physical interventions have suggested promising results. The investigators want to study the effects of our multidisciplinary intensive rehabilitation treatment (MIRT) on balance disorders in PD.

PD patients in stage 3 of Hoen & Yahr will undergo clinical and instrumental evaluations at the beginning (T0) and at the end (T1) of the MIRT. Berg Balance Scale (BBS) will be performed to assess static and dynamic balance abilities. In order to determine some variables as index of postural stability, the investigators will use a stabilometric platform. With respect to the average centre of gravity the standard deviation (SD) of trunk sway will be calculated: total, in antero-posterior (AP) and in medio-lateral (ML) direction. The investigators can obtain a statokinesigram, that is the layout of a line connecting the successive positions of the center of pressure during the recording, and the area of the ellipse containing 90% of the sampled positions of the center of pressure. These measurements will be calculated with open eyes (OE), and while the patient was performing a cognitive task (open eyes counting [OEC]).

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with PD in stage 3 of Hoen & Yahr according to the United Kingdom Brain Bank criteria.

Exclusion criteria:

Atypical parkinsonisms, patients with osteoarticular and muscular pathologies, PD patients with Mini Mental State Examination < 26, patients with other disorders of balance.

Ages: 58 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients (12 M, 18 F, mean age 66,8 ± 8,7) diagnosed with PD in stage 3 of Hoen&Yahr (mean UPDRS III 18.8±10.5) according to the UK Brain Bank criteria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Standard deviation (SD) of trunk sway | up to 4 weeks
  With respect to the average centre of gravity the standard deviation (SD) of trunk sway will be calculated: total, in antero-posterior [AP] and in medio-lateral [ML] direction. We will also calculate a statokinesigram, that is the layout of a line connecting the successive positions of the center of pressure during the recording, and the area of the ellipse containing 90% of the sampled positions of the center of pressure. These measurements will be calculated with open eyes (OE), and while the patient was performing a cognitive task (counting, [OEC]). All physical measurements will be obtained during the ON phase of levodopa medication and at the same time of the day to reduce the influence of medication fluctuations. Statistical analysis with Wilcoxon signed rank test for non parametric data will be performed to analyze differences between T0 and T1 values of all variables. Results will be considered statistically significant for p < 0.05.

SECONDARY OUTCOMES:
BBS scale | up to 4 weeks
  Berg Balance Scale

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Ospedale Generale di Zona "Moriggia-Pelascini", Gravedona ed Uniti (CO), Italy
Locations (1):
- Ospedale Generale di Zona "Moriggia-Pelascini", Gravedona, Como, Italy